CLINICAL TRIAL: NCT06120868
Title: Comparative Clinical Evaluation Between a Novel Self Adhesive and Conventional Bulk-fill Composites (a Randomized Controlled Clinical Study)
Brief Title: Comparative Clinical Evaluation Between a Novel Self Adhesive and Conventional Bulk-fill Composites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 7/2022
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Class II Dental Caries

STUDY DESIGN:
Intervention Model Description: a randomized controlled split-mouth study.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surefil one Self-adhesive bulk fill restorative (SABF) (Experimental)
  Interventions: Other: Surefil one®
- Filtek One Bulk Fill (FOBF) (Active Comparator)
  Interventions: Other: Filtek One

INTERVENTIONS:
Other: Surefil one® — For Surefil one® restorations, the capsule will be activated by pressing it against a stable surface, then mixed in a capsule mixer for 10 s. The capsule tip will be inserted into the proximal box, and the material is extruded as the tip is gradually moved in a coronal direction, ensuring that the material adapts to the cavity bottom and walls.
  Arms: Surefil one Self-adhesive bulk fill restorative (SABF)
Other: Filtek One — Scotchbond™ Universal (SBU) will be used as an adhesive system in self-etch mode for FiltekTM One restoration. SBU will be applied actively for 20 seconds with a disposable brush tip, air-dried gently for 5 seconds to create a consistent bond thickness, then light-cured for 10 seconds. The FiltekTM One will be packed in increments up to 4 mm thick. A second layer of FiltekTM One will be applied on top of the first 4-mm layer if 4 mm is not adequate to properly restore the tooth. Each increment will be light cured for 20 seconds.
  Arms: Filtek One Bulk Fill (FOBF)

SUMMARY:
This study aimed to evaluate the clinical performance of a novel, tooth-colored, self-adhesive bulk-fill restorative, and a conventional bulk-fill composite, for restoring class II cavities.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of restorative treatment on at least two class II Cavities in premolars or molars.
* Presence of proximal caries in digital x-ray with code 2 to 4 according to the radiographic International Caries Detection and Assessment System (ICDAS I).
* Presence of proximal caries in initial or moderate stage according to the International Caries Classification and Management System (ICCMS™).
* Only posterior teeth with class II cavities that have antagonistic contact and at least one proximal contact.
* Absence of parafunctional habits.
* Good general health

Exclusion Criteria:

* Serious medical disorders
* Clinical signs of bruxism, traumatic malocclusion
* Pregnant or breast feeding at the time of restoration placement
* Intolerance or allergy toward the applied restorative materials

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-07-10 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Clinical success of the restoration | up to 12 months
  Clinical success of the restoration will be ranked according to the FDI Clinical Criteria which consider aesthetic, functional, and biological characteristics. The clinical assessment of the investigation criteria will be done by means of a five-score scale. FDI criteria scores 1, 2, and 3 are considered clinically excellent, good, and satisfactory. Score 4 indicates that the restoration is clinically unsatisfactory but repairable, however score 5 indicates that the restoration is clinically poor/failure and should be replaced.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S Ellithy, BDS, Principal Investigator — Alexandria University; Rania R Afifi, PhD, Study Director — Alexandria University; Mohamed H Hussein, PhD, Study Chair — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Derived] Ellithy MS, Abdelrahman MH, Afifi RR. Comparative clinical evaluation between self-adhesive and conventional bulk-fill composites in class II cavities: A 1-year randomized controlled clinical study. J Esthet Restor Dent. 2024 Sep;36(9):1311-1325. doi: 10.1111/jerd.13242. Epub 2024 Apr 24. PMID 38655672